CLINICAL TRIAL: NCT02165371
Title: Sinovuyo Caring Families Project
Brief Title: The Sinovuyo Caring Families Project: a Randomized Controlled Trial of a Parenting Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Oxford (Other); Bangor University (Other)
Responsible Party: Principal Investigator, Dr Catherine L. Ward, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sinovuyo_RCT
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Child Behaviour Problems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sinovuyo Caring Families Programme (Experimental): 12-week group-based parenting program (Sinovuyo Caring Family Programme) delivered in weekly 3 hour sessions. Program is manualized.
  Interventions: Behavioral: Sinovuyo Caring Families Programme
- No intervention (No Intervention): Control group receives not intervention

INTERVENTIONS:
Behavioral: Sinovuyo Caring Families Programme — Goal of the program is reduction in child behavior problems in high-risk South African families. Program will be delivered to caregivers responsible for the wellbeing of the child.
  Program activities will be delivered over 12 weekly group sessions with additional individualized in-home sessions. The groups (n = 15 participants per group) will meet weekly with community facilitators (n = 2 per group). Parenting skills will be developed during the sessions through role-plays, group-discussion, storytelling, and home practice activities.
  The program is manualized in isiXhosa.
  Arms: Sinovuyo Caring Families Programme

SUMMARY:
It has been established that children in families affected by either intimate partner violence or Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome (HIV/AIDS) are at substantially increased risk of poor parenting and child maltreatment. In the sub-Saharan African context of high levels of HIV/AIDS and family violence, it is crucial that parents be supported to establish positive parenting practices and reduce harsh or abusive parenting within their families.This randomized controlled trial will be testing the Sinovuyo Caring Families Program (n = 296), a 12-session (2.5 hour per session) parenting intervention for primary caregivers of children between 2 and 9 years old. Participants will not be restricted to biological parents and include primary caregivers of children between 2 and 9 years old, who live in the same house as the child at least 4 nights per week. Participants will be recruited through systematic household sampling, liaising with Western Cape Department of Social Development and local community-based NGOs. Self-reporting questionnaires and qualitative observational assessment data for intervention and control groups will be collected at pre- and post-test evaluation as well as 12-month follow-up. Primary outcomes will include child behaviour problems, harsh and inconsistent parenting and positive parenting. Secondary outcomes will include parental depression, parental stress, parental monitoring and supervision and parent perceived social support.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver must live with child at least 4 nights per week
* Child must be between 2 and 9 years old Live in Khayelitsha or Nyanga
* May include biological parents, relatives or non-kin foster caregivers, with no restrictions on biological relationship
* Participant must self-identify as the primary caretaker of the child
* Children scoring 15 or higher in the Eyberg Child Behaviour Inventory problem scale

Exclusion Criteria:

* Children scoring 14 or lower in the Eyber Child Behaviour Inventory problem scale
* Participants with child not between 2 and 9 years old
* Participants not self-identifying as the primary care take of the child
* Participants not living with the child at least 4 nights per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory | Baseline, post- intervention and 12-month post-intervention follow-up
  This 36-item examines externalising behaviour problems in children ages 2 to 16 using both an Intensity Scale and Problem Scale. Parents are asked how often a specific behavior occurs and whether the behavior is considered a problem. Based on the most typical child behavior problems, items include "has poor table manners," "acts defiant when told to do something," "physically fights with sisters and brothers," and "fails to finish tasks or project." The Intensity Scale rates frequency of occurrence based on a 7-point Likert scale (1 = never occurs to 7 = always occurs). The Problem Scale measures whether the parent identifies a specific behavior as a problem (0 = no; 1 = yes). Both scales are summed up to create a total Intensity Score and Problem Score. Clinical cut-off scores suggested for psychopathological problem behavior are 131 for the Intensity Score and 11 for the Problem Score (Eyberg, 1999).
Parenting Young Children Scale (Supporting Positive Behaviour subscale; Setting Limits subscale) | Baseline, post- intervention and 12-month post-intervention follow-up
  Parental self-report of positive parenting will be assessed with the Parenting Young Children Scale (PARYC) subscales for supportive positive behaviour and setting limits. The PARYC (21 items total) measures the occurrence of specific parental behaviour towards children during the previous month on a 7-point Likert scale (0 = never; 6 = always), as well as whether performing this behaviour is currently a problem or difficult (0 = no; 1 = yes).
Sinovuyo Observational Coding System | Baseline, post- intervention and 12-month post-intervention follow-up
  This study will also conduct observational assessments of child behaviour using the Sinovuyo Observational Coding System (SOCS). This coding system is based on the Dyadic Parent- Child Interaction Coding System, but has been adapted to be simpler and quicker to use. This tool was developed during the pilot RCT of the Sinovuyo Caring Families Programme to provide a valid and reliable means of coding the behavioural categories that the programme aims to address.

SECONDARY OUTCOMES:
Beck Depression Inventory-II | Baseline, post- intervention and 12-month post-intervention follow-up
  Parental depression will be measured using the Beck Depression Inventory-II (BDI-II). The BDI-II is a 21-item scale with strong psychometric properties and prior use with multiple South African populations.
Parenting Stress Index Short Form | Baseline, post- intervention and 12-month post-intervention follow-up
  Parenting stress will be measured using the Parenting Stress Index (PSI) (36 items). This scale has been used widely throughout the world, including prior use in South African populations. Items are summed to create a total score.
Alabama Parenting Questionnaire (Poor monitoring/supervision subscale) | Baseline, post- intervention and 12-month post-intervention follow-up
  Parental monitoring and supervision will be measured using the Poor Monitoring/Supervision subscale (9 items) of the Alabama Parenting Questionnaire (APQ). Respondents are asked to select how often various actions (e.g., "Your child is home without adult supervision.") have happened in the past month on a 5-point Likert-like scale (1 = never; 5 = always).
Medical Outcome Study Social Support Survey (Emotional Support subscale) | Baseline, post- intervention and 12-month post-intervention follow-up
  Parent perceived social support will be measured using the emotional support subscale of the Medical Outcome Study Social Support Survey (MOS-SSS, 8-items). Parents report on the frequency of how often they receive emotional support (e.g., "someone you can count on to listen to when you need to talk") on a Likert-like scale of 1 to 5 (1 = none of the time; 5 = all of the time). Total scores are calculated by averaging the scores for each item and then transformed into a 0 to 100 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ward, PhD, Principal Investigator — University of Cape Town; Lucie Cluver, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Ikamva Lanbantu Enkululekweni Wellness Centre, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Ward CL, Wessels IM, Lachman JM, Hutchings J, Cluver LD, Kassanjee R, Nhapi R, Little F, Gardner F. Parenting for Lifelong Health for Young Children: a randomized controlled trial of a parenting program in South Africa to prevent harsh parenting and child conduct problems. J Child Psychol Psychiatry. 2020 Apr;61(4):503-512. doi: 10.1111/jcpp.13129. Epub 2019 Sep 19. PMID 31535371